CLINICAL TRIAL: NCT00298233
Title: High-Dose Versus Standard-Dose Oseltamivir for the Treatment of Severe Influenza and Avian Influenza: A Phase II Double-Blind, Randomized Clinical Trial
Brief Title: High-Dose Versus Standard-Dose Oseltamivir to Treat Severe Influenza and Avian Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Wellcome Trust (Other); World Health Organization (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Jeremy Farrar, Director, Oxford University Clinical Research Unit, Oxford University Clinical Research Unit, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SEA 001; N01A050042 (Other Grant/Funding Number: US NIH NIAID Contract)
Record Dates: First submitted 2006-03-01; First posted 2006-03-01 (Estimated); Results first posted 2014-05-22 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Influenza; Avian Influenza; Severe Influenza
Keywords: Antibody Response; Antiviral Efficacy; Bird Flu; Severe Respiratory Distress; Viral Replication and Shedding
MeSH Terms: conditions — Influenza, Human; Influenza in Birds; Dyspnea | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard Dose oseltamivir adult cohort (Active Comparator): All participants >= 15 years will receive standard-dose oseltamivir (75 mg twice daily orally or equivalent dose adjusted for age, weight, and kidney function) for 5 to 10 days.
  Interventions: Drug: Oseltamivir
- Double Dose oseltamivir Adult cohort (Active Comparator): All participants >= 15 years will receive high-dose oseltamivir (150 mg twice daily orally or equivalent dose adjusted for age, weight, and kidney function) for 5 to 10 days.
  Interventions: Drug: Oseltamivir
- Standard Dose Oseltamivir child cohort (Active Comparator): All participants <15 years will receive standard-dose oseltamivir (75 mg twice daily orally or equivalent dose adjusted for age, weight, and kidney function) for 5 to 10 days.
  Interventions: Drug: Oseltamivir
- Double Dose Oseltamivir child cohort (Active Comparator): All Participants <15 years will receive high-dose oseltamivir (150 mg twice daily orally or equivalent dose adjusted for age, weight, and kidney function) for 5 to 10 days.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — Oseltamivir is a sialic acid analogue that potently and specifically inhibits the viral neuraminidases by competitively and reversibly interacting with the active enzyme site of influenza A and B viruses. Oseltamivir will be administered orally in standard formulations (capsules for adults and children at least 15 years of age; suspension for children younger than 15 years).
  Other Names: Tamiflu

SUMMARY:
Influenza, also known as the flu, is a contagious respiratory illness caused by influenza viruses. The illness can range in severity, from mild to severe to even death, and it causes an estimated 500,000 to 1,000,000 deaths worldwide each year. In the last several years, there have been increasing numbers of human cases of avian influenza, or bird flu. This trend may pose a threat of a future pandemic--worldwide outbreak of disease--with an avian influenza virus that can easily spread from person to person. Oseltamivir is an antiviral medication that is used to treat people with uncomplicated human influenza, and it may be effective in treating people with either severe human influenza or avian influenza. The purpose of this international study is to compare standard-dose oseltamivir versus high-dose oseltamivir for treating people who are hospitalized with severe human influenza or avian influenza.

DETAILED DESCRIPTION:
Two main types of influenza virus--Types A and B--are responsible for the seasonal flu epidemics that occur each year. The influenza A viruses can be broken down into subtypes based on two proteins on the surface of the virus: hemagglutinin (H) and neuraminidase (N). The A subtypes usually found in humans are H1N1, H1N2, and H3N2. Other A subtypes are found primarily in animals. For example, the "avian influenza virus" refers to an influenza A virus that is found chiefly in birds.

Although avian influenza does not usually affect humans, increasing numbers of cases of human infection from avian influenza virus H5N1 have been reported in the last several years. Because all influenza viruses have the ability to modify, there is concern that this trend of increasing cases may pose a threat of a future pandemic with a new H5N1 virus that could spread easily from person to person.

The H5N1 virus that has caused human infection in Asia is resistant to amantadine and rimantadine, two antiviral medications commonly used for treating people with influenza. Another antiviral medication, oseltamivir, is currently used to treat people with uncomplicated human influenza. The purpose of this study is to compare standard-dose oseltamivir and high-does oseltamivir for treating people who are hospitalized with severe human influenza or avian influenza. The study will also attempt to identify how severe human influenza and avian influenza differ in the following factors: clinical manifestation, relationship between antiviral plasma concentrations and viral dynamics, and pathogenesis.

Upon meeting certain screening criteria, participants will be randomly assigned to receive oseltamivir either at a standard-dose level (75 mg twice daily orally or equivalent dose adjusted for age, weight, and kidney function) or at a high-dose level (150 mg twice daily orally or equivalent dose adjusted for age, weight, and kidney function). Treatment will continue for 5 days, after which participants who meet clinical failure criteria will continue their assigned treatment for an additional 5 days. It is anticipated that participants will remain hospitalized through the course of treatment. On Day 0, which marks the first day of hospitalization, participants will undergo a medical review, physical examination, blood sampling, nasal swab, throat swab, anal swab, and chest x-ray. An endotracheal aspirate procedure and urine sampling may also be performed. During the hospital stay, most of the above procedures will be repeated regularly, and additional samples of lung fluid, cerebral spinal fluid, and pleural fluid may be obtained. On Day 5 and possibly on Day 10, participants will undergo a follow-up x-ray. If applicable, participants will attend outpatient study visits on Days 10, 14, and 28 for further evaluation; participants with avian influenza will also attend visits on Days 56 and 180.

ELIGIBILITY:
Inclusion Criteria:

* At least one of the following respiratory symptoms: cough, dyspnea, sore throat
* Evidence of severe influenza or avian influenza, as defined below
* Severe influenza infection criteria:

  1. Need for hospitalization
  2. One of the following:

     1. New infiltrate on chest x-ray (or any infiltrate if no prior chest x-ray or not known)
     2. Severe tachypnea (more information on this criterion can be found in the protocol)
     3. Severe dyspnea
     4. Arterial oxygen saturation of 92% or less on room air by trans-cutaneous method
  3. Positive diagnostic testing for influenza, as defined by either rapid influenza antigen (Ag) positive (A or B) or qualitative reverse transcriptase-polymerase chain reaction (RT-PCR) positive for any influenza
  4. Illness (defined by onset of fever, respiratory symptoms, or constitutional symptoms) began within 10 days before study enrollment
* Avian influenza infection criteria:

  1. Nasal wash, nasopharyngeal aspirate, endotracheal aspirate, nasal swab, or throat swab that is RT-PCR positive influenza for H5 influenza
  2. Illness (defined by onset of fever, respiratory symptoms, or constitutional symptoms) began within 14 days before study enrollment

Exclusion Criteria:

* Received more than 72 hours of oseltamivir (six doses) within 14 days
* Received oseltamivir at higher than standard doses within the last 14 days or during current acute illness, whichever is longer
* History of allergy or severe intolerance of oseltamivir, as determined by the investigator
* Alternate explanation for the clinical findings, as determined by the investigator and with the information immediately available
* Creatine clearance less than 10 ml/minute
* Pregnant or breastfeeding

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2006-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tawee Chotpitayasunohdh, MD, Principal Investigator — Queen Sirikit National Institute of Child Health, Bangkok, Thailand; Tran Tinh Hien, MD, Principal Investigator — Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam
Locations (12):
- Singapore (3):
  - Changi General Hospital, Singapore
  - National University Hospital, National University of Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- Thailand (4):
  - Queen Sirikit National Institute of Child Health, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok
  - Bamrasnaradura Infectious Disease Institute, Nonthaburi
  - Chest Disease Institute, Nonthaburi
- Vietnam (5):
  - National Hospital of Pediatrics, Hanoi
  - National Institute fof Infectious and Tropical Diseases, Hanoi
  - Children's Hospital #1, Ho Chi Minh City
  - Hospital for Tropical Diseases, Ho Chi Minh City
  - Pediatric Hospital #2, Ho Chi Minh City

REFERENCES:
- [Background] Morse SS. Factors in the emergence of infectious diseases. Emerg Infect Dis. 1995 Jan-Mar;1(1):7-15. doi: 10.3201/eid0101.950102. PMID 8903148
- [Background] Colman PM. Influenza virus neuraminidase: structure, antibodies, and inhibitors. Protein Sci. 1994 Oct;3(10):1687-96. doi: 10.1002/pro.5560031007. PMID 7849585
- [Background] de Jong MD, Bach VC, Phan TQ, Vo MH, Tran TT, Nguyen BH, Beld M, Le TP, Truong HK, Nguyen VV, Tran TH, Do QH, Farrar J. Fatal avian influenza A (H5N1) in a child presenting with diarrhea followed by coma. N Engl J Med. 2005 Feb 17;352(7):686-91. doi: 10.1056/NEJMoa044307. PMID 15716562
- [Result] South East Asia Infectious Disease Clinical Research Network. Effect of double dose oseltamivir on clinical and virological outcomes in children and adults admitted to hospital with severe influenza: double blind randomised controlled trial. BMJ. 2013 May 30;346:f3039. doi: 10.1136/bmj.f3039. PMID 23723457

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Dose Oseltamivir Adult Cohort: All participants >= 15 years received standard-dose oseltamivir (75 mg twice daily orally or equivalent dose adjusted for age, weight, and kidney function) for 5 to 10 days.
- Double Dose Oseltamivir Adult Cohort: All Participants >= 15 years received high-dose oseltamivir (150 mg twice daily orally or equivalent dose adjusted for age, weight, and kidney function) for 5 to 10 days.
- Standard Dose Oseltamivir Child Cohort: All participants <15 years received standard dose oseltamivir (75 mg twice daily orally or equivalent dose adjusted for age, weight, and kidney function) for 5 to 10 days.
- Double Dose Oseltamivir Child Cohort: All Participants <15 years received high-dose oseltamivir (150 mg twice daily orally or equivalent dose adjusted for age, weight, and kidney function) for 5 to 10 days.
Period: Overall Study
Arm/Group | Standard Dose Oseltamivir Adult Cohort | Double Dose Oseltamivir Adult Cohort | Standard Dose Oseltamivir Child Cohort | Double Dose Oseltamivir Child Cohort
Started | 39 | 41 | 122 | 124
Completed | 39 | 41 | 122 | 124
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants that were randomized
Groups:
- Standarad Dose Oseltamivir: All participants that were randomized and received standard dose oseltamivir
- Double Dose Oseltamivir: All participants that were randomized and received doubledose oseltamivir
- Total: Total of all reporting groups
Arm/Group | Standarad Dose Oseltamivir | Double Dose Oseltamivir | Total
Number analyzed (Participants) | 161 | 165 | 326
Age, Customized [Number; unit: participants]
  Child cohort: ≥1 to <15 years | 122 | 124 | 246
  Adult cohort: ≥15 years | 39 | 41 | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 69 | 141
  Male | 89 | 96 | 185

OUTCOME MEASURES:

1. Primary Outcome: Proportion of All Participants Negative for Viral RNA on Day 5
Description: Proportion of all participants with no detectable viral RNA by reverse transcriptase-polymerase chain reaction (RT-PCR) in a combined nasal and throat swab sample on day 5.
Time Frame: After 5 days of treatment
Population: All randomized patients with RT-PCR proven influenza.
Measure: Number; unit: participants
Groups:
- Double Dose Oseltamivir: All participants receiving double dose oseltamivir
- Standard Dose Oseltamivir: All participants receiving standard dose oseltamivir
Arm/Group | Double Dose Oseltamivir | Standard Dose Oseltamivir
Number analyzed (Participants) | 159 | 154
participants | 115 | 105
Statistical Analysis 1: Comparison: Double Dose Oseltamivir vs Standard Dose Oseltamivir; Based on previous studies, assumption was made that 30% of children and 55% of adults treated with standard dose oseltamivir would test negative for virus on day five. This would require a sample size of 242 patients to show a 20% absolute improvement in cessation of viral shedding with 85% power and a two sided α of 0.05. To allow for study withdrawals, the target sample size was set at 300 patients; Test type: Superiority or Other; p = 0.42, conditional univariate logistic regressi — Significance assessed at the 5% level for a two-sided comparison; analysis stratified by study site

2. Secondary Outcome: Participants Meeting Criteria for Day 5 Clinical Failure
Description: Proportion of participants that have clinical failure by day 5. Subjects that meet one of the following on Day 5 will be classified as a clinical failure:
  * Severe tachypnea (respiratory rate ≥ 30 for ages ≥12 years, rate ≥ 40 for ages 6 to 12 years, rate ≥45 for ages 3 to 6 years, rate ≥ 50 for ages 1 to 3 years)
  * Severe dyspnea (unable to speak full sentences, or use of accessory respiratory muscles)
  * Arterial oxygen saturation ≤92% on room air by trans-cutaneous method
  * Need for mechanical ventilation or intensive care unit (ICU) admission For the purpose of endpoint definition, death prior to or on Day 5 will also be considered a clinical failure at Day 5.
Time Frame: After 5 days of treatment
Population: For the purpose of endpoint definition, death prior to or on Day 5 was also considered as clinical failure on day 5.In the double dose cohort, only 154 subjects completed fives days of drug and 7 died (total 161). In the standard dose cohort only 149 subjects completed 5 days of drug and 9 died (total 158).
Measure: Number; unit: participants
Arm/Group | Double Dose Oseltamivir | Standard Dose Oseltamivir
Number analyzed (Participants) | 161 | 158
participants | 16 | 20
Statistical Analysis 1: Comparison: Double Dose Oseltamivir vs Standard Dose Oseltamivir; Test type: Superiority or Other; p = 0.54, Mantel Haenszel — Significance assessed at the 5% level for a two-sided comparison

3. Secondary Outcome: In-hospital Mortality Rates
Description: Standard therapy with oseltamivir is five days. Those patients with persistent symptoms on day five were continued on the randomized dose for an additional five days and assessments were performed up to day 10.
Time Frame: After up to 10 days of treatment
Measure: Number; unit: participants
Arm/Group | Double Dose Oseltamivir | Standard Dose Oseltamivir
Number analyzed (Participants) | 165 | 161
participants | 12 | 9
Statistical Analysis 1: Comparison: Double Dose Oseltamivir vs Standard Dose Oseltamivir; Test type: Superiority or Other; p = 0.54, Mantel Haenszel — Significance assessed at the 5% level for a two-sided comparison; Mantel-Haenszel chi-square stratified by study site

4. Secondary Outcome: Median Time (Days) Receipt of Oxygen
Time Frame: Throughout study, 14 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Double Dose Oseltamivir | Standard Dose Oseltamivir
Number analyzed (Participants) | 165 | 161
days | 3 (2-5) [2 to 5] | 3.5 (2-7) [2 to 7]
Statistical Analysis 1: Comparison: Double Dose Oseltamivir vs Standard Dose Oseltamivir; Test type: Superiority or Other; p = 0.48, Kruskal-Wallis — Significance assessed at the 5% level for a two-sided comparison

5. Secondary Outcome: Median Time (Days) in ICU
Time Frame: Throughout study, 14 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Double Dose Oseltamivir | Standard Dose Oseltamivir
Number analyzed (Participants) | 165 | 161
days | 4.4 [3 to 6] | 5 [2 to 11]
Statistical Analysis 1: Comparison: Double Dose Oseltamivir vs Standard Dose Oseltamivir; Test type: Superiority or Other; p = 0.66, Kruskal-Wallis — Significance assessed at the 5% level for a two-sided comparison

6. Secondary Outcome: Median Time (Days) on Ventilation
Description: Use of mechanical ventilation at any time for subjects with severe influenza and avian influenza.
Time Frame: Throughout study, 14 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Double Dose Oseltamivir | Standard Dose Oseltamivir
Number analyzed (Participants) | 165 | 161
days | 2.5 [1 to 16] | 5 [2 to 11]
Statistical Analysis 1: Comparison: Double Dose Oseltamivir vs Standard Dose Oseltamivir; Test type: Superiority or Other; p = 0.58, Kruskal-Wallis — Significance assessed at the 5% level for a two-sided comparison

ADVERSE EVENTS:
Time Frame: Through Day 28 for severe influenza, and Day 180 for avian influenza.
Description: The study recorded only cumulative data (total number of AEs per type, per Arm, but not number of subjects affected per AE type). Therefore data are the number of events and not the number of participants with events.
Groups:
- Double Dose Oseltamivir; Standard Dose Oseltamivir: The study recorded only cumulative data (total number of adverse events (AEs) per type, per Arm, but not number of subjects affected per AE type). Therefore data are the number of events and not the number of participants with events.
Arm/Group | Double Dose Oseltamivir | Standard Dose Oseltamivir
Serious Adverse Events (participants affected / at risk) | 1/165 | 0/161
Other Adverse Events (participants affected / at risk) | 37/165 | 38/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Dose Oseltamivir (N=165) | Standard Dose Oseltamivir (N=161)
Septic shock (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — A participant was admitted to the hospital for suspected pneumonia. Following upper GI bleeding and respiratory failure, diagnosis confirmed as septic shock. Subject eventually stabilized. Unblinding revealed subject was on high dose oseltamivir.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Dose Oseltamivir (N=165) | Standard Dose Oseltamivir (N=161)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 5 (5)
diarrhea (Gastrointestinal disorders) | 2 (2) | 9 (9)
multi-organ failures (General disorders) | 3 (3) | 3 (3)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Septic shock (Cardiac disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
other (General disorders) | 10 (10) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No